CLINICAL TRIAL: NCT01826799
Title: Noise in the Intensive Care Unit and Its Influence on Sleep Quality: a Nationwide Survey in Dutch Intensive Care Units
Brief Title: Noise in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, K.S. Simons, MD, Jeroen Bosch Ziekenhuis
Other Study IDs: ICUnoise
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Noise in the ICU; Sleep Quality in Adult ICU Patients
Keywords: sleep; noise; ICU; delirium; RCSQ
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- adult ICU patients: All adult patients without hearing disabilities and admitted to the ICU more than 48 hours ago, with a Richmond Agitation-Sedation Scale (RASS) of -2 or higher and the capability to understand Dutch are eligible.

SUMMARY:
Rationale: Sound levels in the Intensive Care Unit are frequently reported to exceed the recommended levels. It is plausible to assume that this causes sleep disturbance in the patients on the ICU.

Goals/endpoints: to assess sound pressure levels in 6 different Dutch ICU´s and evaluate the effect of higher levels on sleep as perceived by the patient.

Study design: observational multicenter study

Study population: adult ICU patients > 18 years old with an expected duration of stay of more than 24 hours

Study parameters/endpoints:

Primary

1. To gather information on how Dutch ICUs perform on sound levels

   1. Average sound pressure level
   2. Number of sound peaks
2. To question patients about their perception of sleep quality (measured by RCSQ)
3. Causes of elevated sound pressure levels
4. Identification of the most annoying sounds experienced by the patient

Secondary

1) Incidence of delirium measured by CAM-ICU

DETAILED DESCRIPTION:
An exploratory prospective-observational multi-center study with a total of 6 participating hospitals will be performed. We will include 15 patients per center. Characteristics of the participating ICUs will be collected.All adult patients without hearing disabilities and admitted to the ICU more than 48 hours ago, with a Richmond Agitation-Sedation Scale (RASS) of -2 or higher and the capability to understand Dutch are eligible.Sound measurement equipment will be installed in two patient rooms in each ICU and will perform a continuous recording. Sound parameters that will be measured include average sound levels, number and height of peaks and peak-to-baseline level.

Level of sedation is monitored as part of daily care by nurses in all patients every two hours using the RASS.In addition, screening on the presence of delirium is done using the Confusion Assessment Method-ICU (CAM-ICU) every shift.Patients' perception of sleep will be scored (both by the patient and the attending nurse) using the Richards-Campbell Sleep Questionnaire (RCSQ),after the 24 hour recording period from the start of the inclusion and from there on every 24 hours until discharge with a maximum of five days at 07.00 am by the attending nurse.

Data, consisting of patient information and results of measurements and laboratory investigations will be filled in on an electronic Case Record Form (e-CRF).

For the descriptive statistics, values will be given as mean ± SD or median and interquartile ranges, depending on their distribution. Summary tables will be provided for all baseline and follow-up variables. Data will be summarised by producing frequently tabulations for categorical variables and summary statistics for continuously distributed variables with confidence intervals.

All statistical tests are two-sided and statistical significance is defined as a P-value <0.05. All data are analyzed using SPSS version 18.0 (SPSS, Chicago, IL).

Association between noise and delirium will be evaluated using a logistic multivariate regression analysis, correcting for age, severity of disease, infection and sedative use

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patient
* RASS -2 - +1

  * 48 hours after admission on ICU
* Expected ICU stay >24 hours

Exclusion Criteria:

* Unfavourable prognosis (life expectancy < 48 hours)
* Inability to understand Dutch, including total deafness
* Inability to complete visual analog scale due to visual impairment blindness, and/or severe psychomotor retardation
* Delirium (defined as positive CAM-ICU)
* Participation of the patient in other studies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients without hearing disabilities and admitted to the ICU more than 48 hours ago, with a Richmond Agitation-Sedation Scale (RASS) of -2 or higher and the capability to understand Dutch are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Noise Level | 6 months
  To gather information on how Dutch ICUs perform on sound levels
  1. Average sound pressure level (e.g. per shift, over day/night)
  2. Number of sound peaks
  3. Peak-to-baseline level
  4. Etiology of noise - classification of dominant sources

SECONDARY OUTCOMES:
Sleep quality of ICU patients | 6 months
  Patients' perception of sleep will be scored (both by the patient and the attending nurse) using the Richards-Campbell Sleep Questionnaire (RCSQ, see appendix). This will take place after the 24 hour recording period from the start of the inclusion and from there on every 24 hours until discharge with a maximum of five days at 07.00 am by the attending nurse. An additional question will be added to the RCSQ, namely which sound the patient has experienced to be the most annoying/disturbing during his/her stay in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Simons, MD, Principal Investigator — Jeroen Bosch Ziekenhuis
Locations (6):
- Netherlands (6):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Elisabeth Ziekenhuis, Tilburg, North Brabant
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel

REFERENCES:
- [Derived] Simons KS, Verweij E, Lemmens PMC, Jelfs S, Park M, Spronk PE, Sonneveld JPC, Feijen HM, van der Steen MS, Kohlrausch AG, van den Boogaard M, de Jager CPC. Noise in the intensive care unit and its influence on sleep quality: a multicenter observational study in Dutch intensive care units. Crit Care. 2018 Oct 5;22(1):250. doi: 10.1186/s13054-018-2182-y. PMID 30290829